CLINICAL TRIAL: NCT07124312
Title: Placental Characteristics Within Monochorionic Twin Pregnancies: a Prospective Cohort Study.
Brief Title: Placental Characteristics Within Monochorionic Twin Pregnancies
Status: Recruiting | Type: Observational
Sponsor: Birmingham Women's NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Jack Hamer, Clinical research fellow, Birmingham Women's NHS Foundation Trust
Other Study IDs: 24/BW/MAT/NO/852
Record Dates: First submitted 2025-08-01; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Placenta; Monochorionic Twins; Anatomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uncomplicated monochorionic twins: Monochorionic twins which do not develop any complications during the antenatal period
- Complicated monochorionic twins: Monochorionic twins which develop any type of complication during the antenatal period such as TTTS, sIUGR and TAPS.

SUMMARY:
This prospective study aims to collate a comprehensive database of all main monochorionic twin groups to enable comparisons to be made within each twin group and additionally between each group with regards to several placental characteristics, whilst understanding their impact on several fetal outcomes. This study aims to provide new insights in to how the placental architecture influences pregnancy care within the UK pregnancy cohort. Results of this study may impact how clinicians conduct antenatal surveillance for these anatomical placental factors.

Patients of both uncomplicated and complication monochorionic twin groups will be consented at a single site and recruited during the antenatal period. Following delivery the placenta will then be analysed macroscopically and assessed for several anatomical features. This will be compared with the antenatal complications and perinatal outcomes for the respective twin.

ELIGIBILITY:
Inclusion Criteria:

• All consecutive placentas of monochorionic twin pregnancies whereby the placenta is transferred to the pathology department for analysis.

Exclusion Criteria:

* Singleton, dichorionic and higher order pregnancies (e.g. triplet).
* Fetus with known major congenital anomalies or aneuploidy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Placentas received within the pathology department from monochorionic twin groups . These groups include:
  * Uncomplicated monochorionic twins
  * Monochorionic twins with complications (e.g. selective intrauterine growth restriction, twin-twin transfusion syndrome , twin anaemia-polycythaemia sequence etc).
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
What is the impact of intertwin vascular anastomoses on fetal complications and perinatal outcome | Throughout the study period (approximately 2 years)
  To determine the prevalence of intertwin vascular anastomoses (overall, artery-artery, artery-vein, vein-vein) on adverse perinatal outcome (e.g. stillbirth and neonatal death) and fetal complications (e.g. small for gestational age). Measures will be as overall percentages and also raw numbers which will be calculated in to odds ratio's when comparing anastomoses versus no anastomoses against the respective perinatal outcome and fetal complication
What is the impact of abnormal cord insertion on fetal complications and perinatal perinatal outcome | Throughout the study period (approximately 2 years
  To determine the prevalence of abnormal cord insertion (marginal and velamentous) on adverse perinatal outcome (e.g. stillbirth and neonatal death) and fetal complications (e.g. small for gestational age, selective growth restriction). Measures will be as overall percentages and also raw numbers which will be calculated in to odds ratio's when comparing abnormal cord insertion versus normal cord insertion against the respective perinatal outcome and fetal complication
What is the impact of twin placental sharing on fetal complications and perinatal outcome | Throughout the study period (approximately 2 years)
  To determine the impact of placental sharing between each twin on adverse perinatal outcome (e.g. stillbirth and neonatal death) and fetal complications (e.g. birthweight discordance and selective growth restriction). Placental sharing will be defined as a percentage of overall share between each twin which sums up to 100%. The difference between each twin's share will be determine by minimising the larger percentage from the smaller percentage. The difference will then be compared to adverse perinatal outcomes and complications such as selective growth restriction using odds ratio's. Birthweight discordance will be defined as a percentage ( difference between the larger twin weight and smaller twin weight, divided by the larger twin weight). This will be compared to placental sharing using a graphical comparison of all placental sharing results, individually compared against each respective birthweight discordance.

SECONDARY OUTCOMES:
The influence of abnormal cord insertion in monochorionic twins complicated by twin-twin transfusion syndrome | Throughout the study period (approximately 2 years)
  To understand the frequency of abnormal cord insertion (marginal and velamentous) within monochorionic twins complicated by twin-twin transfusion syndrome following laser ablation and determine the impact on fetal outcomes such as stillbirth, neonatal death, recurrent twin-twin transfusion syndrome and twin anaemia-polycythaemia sequence. Results will be collected as overall number of placentas with abnormal cord (both marginal, velamentous and both) and those with normal cord insertion, and compared against the number of events in the respective fetal outcome. Results will be presented as odds ratio's.
The influence of residual vascular anastomoses monochorionic twins complicated by twin-twin transfusion syndrome | Throughout the study period (approximately 2 years)
  To understand the frequency of residual vascular anastomoses within monochorionic twins complicated by twin-twin transfusion syndrome following laser ablation and determine their impact on fetal outcomes such as stillbirth, neonatal death, recurrent twin-twin transfusion syndrome and twin anaemia-polycythaemia sequence. Results will be collected as overall number of placentas with residual vascular anastomoses, alongside the individual types of anastomoses (artery-artery, artery-vein, vein-vein) and compared against the number of events in the respective fetal outcome. Results will be presented as odds ratio's.
The influence of abnormal cord insertion on residual anastomoses development in monochorionic twins complicated by twin-twin transfusion syndrome undergoing laser ablation | Throughout the study period (approximately 2 years)
  To understand the impact of abnormal cord insertion (marginal and velamentous) on residual anastomoses development in monochorionic twins complicated by twin-twin transfusion syndrome undergoing laser ablation. Results will be collected as overall number of placentas with abnormal cord insertion and whether they have residual anastomoses versus those without abnormal cord insertion and if they have residual anastomoses seen. Results will be presented as odds ratio's.
Examine the association between Quintero staging during laser ablation for monochorionic twins complicated by twin-twin transfusion syndrome on residual anastomoses development | Throughout the study period (approximately 2 years)
  To examine the impact of Quintero staging during laser ablation for twin-twin transfusion syndrome on the frequency of post-laser residual anastomoses. Quintero staging will be split in to the four stages and expressed as overall numbers versus the number of placentas with and without residual anastomoses. Results will be expressed as odds ratio's.
Examine the relationship between placenta position during laser ablation for monochorionic twins complicated by twin-twin transfusion syndrome and the rate of residual anastomoses development. | Throughout the study period (approximately 2 years)
  To examine the impact of placenta position during laser ablation for twin-twin transfusion syndrome on the frequency of post-laser residual anastomoses. Placenta position will be either anterior or posterior and expressed as overall numbers versus the number of placentas with and without residual anastomoses. Results will be expressed as odds ratio's.
The influence of intertwin cord distance on fetal complications | Throughout the study period (approximately 2 years)
  The assess the intercord twin distance on fetal complications such birthweight discordance. The distance of the twin cords will be measured in centimetres. This distance will be divided by the distance of the overall placental length to form a number between 0-1. This will then be compared graphically against birthweight discordance, which will be presented as a percentage (difference between the larger twin weight and smaller twin weight, divided by the larger twin weight).
Determine the frequency of abnormal cord insertion in monochorionic twin groups | Throughout the study period (approximately 2 years)
  To determine the frequencies of abnormal cord insertion (velamentous and marginal) in monochorionic twin groups. This will be defined as percentages (number of cases with abnormal cord (velamentous, marginal and both) divided by the overall number) in each twin group (uncomplicated, twin-twin transfusion, selective growth restriction, twin anaemia-polycythaemia, TRAP, monoamniotic). Results will be compared to each group using P values.
Determine the frequency of intertwin anastomoses in monochorionic twin groups | Throughout the study period (approximately 2 years)
  To determine the frequencies of intertwin vascular anastomoses (overall, artery-artery, artery-vein, vein-vein) in monochorionic twin groups. This will be defined as percentages (number of cases with intertwin vascular anastomoses (overall, artery-artery, artery-vein, vein-vein) divided by the overall number in each twin group (uncomplicated, twin-twin transfusion, selective growth restriction, twin anaemia-polycythaemia, TRAP, monoamniotic). Results will be compared to each group using P values

CONTACTS AND LOCATIONS:
Overall Officials: Jack Hamer, MBChB, Principal Investigator — Birmingham Women's and Children's NHS Foundation Trust
Locations (1):
- Birmingham Women's and Children's NHS Foundation Trust, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No